CLINICAL TRIAL: NCT03301155
Title: International Multicenter Double-bind Placebo-controlled Randomized Parallel-group Clinical Trial of Anaferon for Children Efficacy in Prevention of Influenza and Other Acute Respiratory Viral Infections in Children During the Peaks of Seasonal Morbidity
Brief Title: Clinical Trial of Anaferon for Children Efficacy in Prevention of Influenza and Other ARVI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MMH-AD-008
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Results first posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2019-05

CONDITIONS: Preventive Medicine
MeSH Terms: interventions — anaferon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anaferon for children (Experimental): Tablet for oral use. One tablet per intake, once daily (approximately at the same time).
  The product is administered outside a meal (in the interval between meals or 15 min prior to meal or fluid intake), the tablets should be held in mouth until complete dissolution. For young children (aged 1 month to 3 years old), the tablet is recommended to be dissolved in a small amount (1 tablespoon) of drinking water of room temperature.
  Interventions: Drug: Anaferon for children
- Placebo (Placebo Comparator): Tablet for oral use. Placebo using Anaferon for children scheme.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anaferon for children — Tablet for oral use.
  Arms: Anaferon for children
Drug: Placebo — Tablet for oral use.
  Arms: Placebo

SUMMARY:
The objective of this study is to obtain additional data on the efficacy and safety of 12-week course of therapy with Anaferon for children for prevention of influenza and other acute respiratory viral infections in children during the peaks of seasonal morbidity.

DETAILED DESCRIPTION:
Design: an international, multicenter, double-blind, placebo-controlled, randomized study in parallel groups.

The study will enroll children of either gender aged of 1 month to 6 years old. Children can participate in the study, regardless of the frequency of previous ARVI. A potential study participant should not be in the incubation (if known), prodromal, acute/subacute periods of any infectious disease (except for the recovery period). Schedule for enrollment of participants: during the period of a seasonal rise in influenza/ARVI incidence in the Russian Federation and the Republic of Uzbekistan. Screening and randomization of participants will be subject to availability of official information on the incidence of influenza/ARVI in the relevant study region.

The doctor makes the first visit to the participant in the medical center or at home. After the parent/adoptive parent signs the information sheet (informed consent form), the doctor evaluates the possibility of the participant being included in the trial. If the child meets all the inclusion criteria and does not have all non-inclusion criteria, then he/she is included in the study, the doctor fills in Clinical Research Form. At visit 1 (Day 1), the participant is randomized into one of two groups: the 1st group participants will take Anaferon for children according to the preventive regimen for 12 weeks; the 2nd group participants will take Placebo according to the regimen of Anaferon for 12 weeks.

In total, the study participant will be observed for 12 weeks (screening and randomization up to 1 day, preventive treatment for 12 weeks).

During the observation period at 4 (Visit 2), 8 (Visit 3) and 12 (Visit 4) weeks, three visits are planned.

Visits 2 (Week 4 ± 3 days) and 3 (Week 8 ± 3 days) are conducted in the form of a telephone survey of parents/adoptive parents about the participant's health status, presence/absence of symptoms of influenza/ARVI, possible use of antibacterial drugs and/or hospitalization during the course preventive therapy.

Visit 4 (Week 12 ± 3 days) is carried out at home or in a medical center; the doctor collects complaints, examines the participant, registers concomitant therapy, assesses the compliance of the therapy.

If in the period from 2 to 12 weeks a participant falls ill with influenza/ARVI, then he/she prematurely completes participation in the study (as having reached the primary endpoint). A participant is considered fallen ill with influenza/ARVI if the doctor identifies the following symptoms: febrile/subfebrile body temperature, presence at least one flu-like nonspecific symptom (decreased activity/impaired behavior/weakness; headache; chills) and at least one respiratory symptom (runny nose; nasal stuffiness; hoarseness/husky voice; sore throat; cough). In this case, the doctor makes an unscheduled visit (at home or in a medical center), which is final. During the visit, the doctor carries out the procedures of Visit 4. A nasopharyngeal swab is taken to identify the most common pathogens of influenza/ARVI.

If ARVI/influenza occurs within the first seven days from the onset of preventive therapy, the disease will not be recorded as an adverse event and will not be taken into account to evaluate the efficacy of the study drug, since an early manifestation of influenza/ARVI may indicate that the participant was included in the study when he/she was in the incubation period of an infectious disease.

During the study, concomitant therapy for underlying chronic conditions, as well as routine vaccination of the participant, are allowed, with the exception of the drugs indicated in the section "Prohibited Concomitant Treatment".

ELIGIBILITY:
Inclusion Criteria:

1. Children of either gender aged from 1 month to 6 years old.
2. The absence of clinical symptoms of any infectious disease, but not earlier than 14 days from its onset.
3. Seasonal rise in ARVI incidence, confirmed by official information.
4. An information sheet (Informed Consent form) for the subject participation in the clinical trial signed by one parent/adopter of the patient.

Exclusion Criteria:

1. Acute or subacute period of infectious disease of any etiology (viral, bacterial, fungal, etc.) and localization (including upper and lower respiratory tract infection, meningitis, sepsis, otitis media, urinary tract infection, intestinal infection, etc.).
2. History of (verified previously) or current suspected conditions such as:

   * primary or secondary immunodeficiency;
   * bronchopulmonary dysplasia, primary ciliary dyskinesia, cystic fibrosis, other chronic pulmonary diseases;
   * malformations of the respiratory and ENT organs (ear, throat, mouth, tongue, larynx, trachea, neck and salivary and thyroid glands, etc.);
   * immunopathological diseases (including Marshall syndrome, Behсet's syndrome, Kawasaki disease, etc.);
   * hematological diseases (including agranulocytosis, leukemia);
   * oncologic conditions.
3. Exacerbated or decompensated of chronic diseases affecting the patienrt's ability to participate in the clinical trial.
4. Malabsorption syndrome, including congenital or acquired lactase or another disaccharide deficiency, galactosemia.
5. Allergy/intolerance to any component of the study drug.
6. Course administration of the drug products specified in the section 'Prohibited concomitant medications' within 2 weeks prior to enrollment.
7. Children whose parents/adopter parents will fail to comply with the observation requirements of the trial or with the intake regimen of the study drug, from the investigator's point of view.
8. Participation in other clinical trials within 3 month prior to enrollment in the study.
9. The patient's parent/adopter parent is a member of the research team of the investigational site directly involved in the study or a close relative of an investigator. Close relatives are defined as husband/wife, parents, children, brothers (sisters) regardless of whether they are biological or adopted.
10. The patient's parent/adopter parent works for OOO "NPF "MATERIA MEDICA HOLDING" (i.e., the company's employee, part-time employee under contract or appointed official in charge of the trial, or their immediate family).

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1036 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- Russia (32):
  - Regional budgetary health care institution "Regional Children's Clinical Hospital", Ivanovo
  - Republican Children's Clinical Hospital of the Ministry of Health of the Udmurt Republic, Izhevsk
  - Federal State Budgetary Educational Institution of Higher Education "Kazan Medical University" of the Ministry of Healthcare of the Russian Federation, Kazan'
  - Kazan Federal University, Kazan'
  - Federal Budget Institution of Science "Central Research Institute of Epidemiology" of The Federal Service on Customers' Rights Protection and Human Well-being Surveillance, Moscow
  - Federal State Budgetary Educational Institution of Higher Education "Pirogov Russian National Research Medical University" of the Ministry of Healthcare of the Russian Federation, Moscow
  - State Federal-Funded Educational Institution of Higher Professional Training I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation, Moscow
  - LLC Center for Vaccine Prevention "DIAVAKS", Moscow
  - Limited Liability Company "Gubernskiy lekar'", Murmansk
  - Limited Liability Company "MDP-Medical Group", Odintsovo
  - Federal State Budgetary Educational Institution of Higher Education "Orenburg State Medical University" of the Ministry of Healthcare of the Russian Federation, Orenburg
  - Municipal Health Care Institution "City Child Health Clinical Polyclinic №5", Perm
  - Municipal Budgetary Health Care Institutions "Semashko City Hospital №1 Rostov-on-Don ", Rostov-on-Don
  - Municipal budgetary health care institution "Children's city polyclinic №4", Rostov-on-Don
  - St. Petersburg State Budgetary Healthcare Institution "Children's City Polyclinic No. 44", Saint Petersburg
  - St. Petersburg State Budgetary Health Care Institution "Сity Polyclinic №44", Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "St. Petersburg State Pediatric Medical Academy" of Ministry of Health of Russian Federation, Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "Children's City Polyclinic No. 35", Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "Children's City Hospital No. 22", Saint Petersburg
  - Samara Regional Children's Sanatorium "Yunost'", Samara
  - State Budgetary Institution of Health of the Samara Region "Samara City Children's Clinical Hospital No. 1 named after N.N. Ivanova", Samara
  - Limited Liability Company "DNA Research Center", Saratov
  - Regional State Autonomous Healthcare Institution "Children's Hospital №1", Tomsk
  - Siberian State Medical University, Tomsk
  - Bashkir State Medical University, Ufa
  - Volgograd State Medical University/Departmental Clinical Hospital at Volgograd-1 Station of Russian Railways, Volgograd
  - Volgograd State Medical University/Volgograd Regional Clinical Hospital # 1, Volgograd
  - Yaroslavl State Medical University/Children's Clinic # 5, Yaroslavl
  - Yaroslavl State Medical University/Clinical Hospital # 8 (Children's Clinic # 1), Yaroslavl
  - Yaroslavl State Medical University/Department of Infectious Diseases, Epidemiology and Children's Diseases, Yaroslavl
  - Yaroslavl State Medical University/Regional Children's Clinical Hospital # 8 (Children's Clinic # 2), Yaroslavl
  - Municipal Autonomous Institution "Children's City Clinical Hospital No. 11", Yekaterinburg
- Family polyclinic № 6, Tashkent, Uzbekistan

RESULTS

PARTICIPANT FLOW:
Groups:
- Anaferon for Children: Tablet for oral use. One tablet per intake, once daily (approximately at the same time).
  The product is administered outside a meal (in the interval between meals or 15 min prior to meal or fluid intake), the tablets should be held in mouth until complete dissolution. For young children (aged 1 month to 3 years old), the tablet is recommended to be dissolved in a small amount (1 tablespoon) of drinking water of room temperature.
  Anaferon for children: Tablet for oral use.
Period: Overall Study
Arm/Group | Anaferon for Children | Placebo
Started | 528 | 508
Completed | 520 | 501
Not Completed | 8 | 7
Not completed — Сompliance with exclusion criteria | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anaferon for Children | Placebo | Total
Number analyzed (Participants) | 520 | 501 | 1021
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 520 | 501 | 1021
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.1 (1.7) | 3.1 (1.7) | 3.1 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263 | 244 | 507
  Male | 257 | 257 | 514
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Uzbekistan | 15 | 15 | 30
  Russia | 505 | 486 | 991

OUTCOME MEASURES:

1. Primary Outcome: Time From Taking the First Dose of the Study Drug to the Onset of Influenza/ARVI Symptoms.
Description: Based on medical records.
Time Frame: in 12 weeks of the treatment
Population: Intention-to-treat (ITT)
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 520 | 501
days | 428.8 [351.0 to 523.8] | 275.8 [232.7 to 326.9]
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p = 0.001, Regression, Logistic; Comparison performed on the regression parameters scale. Estimates for mean time obtained under assumption of exponentially distributed time-to-event
Statistical Analysis 2: Comparison: Anaferon for Children vs Placebo; Test type: Superiority — superiority margin for hazard ratio was prespecified as 0.846. Lower hazard is better thus the upper confidence limit of HR expected to be lesser than margin; p = 0.0218, Regression, Cox; Hazard Ratio (HR) = 0.645, 95% CI 2-sided [0.496 to 0.839] — Lower HR is better

2. Secondary Outcome: Percentage of Children Not Falling Ill With Influenza or Another ARVI.
Description: Based on medical records. Influenza/ARVI criteria are the following: febrile/subfebrile body temperature, presence at least one flu-like nonspecific symptom (decreased activity/weakness, headache, and chills), and at least one respiratory symptom (runny nose, nasal stuffiness, hoarseness/husky voice, sore throat, and cough).
Time Frame: in 12 weeks of the treatment
Population: Intention-to-treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 520 | 501
Participants
  4 weeks | 516 | 452
  8 weeks | 482 | 415
  12 weeks | 424 | 368
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Comparison between groups on week 4; Test type: Superiority; p = 0.0003, Fisher Exact — Adjusted with Holm method for multiple comparrisons
Statistical Analysis 2: Comparison: Anaferon for Children vs Placebo; Comparison between groups on week 8; Test type: Superiority — Adjusted with Holm method for multiple comparrisons; p = 0.0003, Fisher Exact
Statistical Analysis 3: Comparison: Anaferon for Children vs Placebo; Comparison between groups on week 12; Test type: Superiority; p = 0.0021, Fisher Exact

3. Secondary Outcome: Percentage of Children With the Symptoms Requiring Antibacterial Therapy.
Description: Based on medical records. Percentage of children with the symptoms of a respiratory or ear-nose-throat bacterial infection requiring antibacterial therapy.
Time Frame: in 12 weeks of the treatment
Population: Intention-to-treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 520 | 501
Participants | 3 | 8
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p = 0.1372, Fisher Exact

4. Secondary Outcome: Percentage of Children Requiring Hospitalized for Influenza/ARVI.
Description: Based on medical records. Percentage of children hospitalized for influenza/ARVI or their complications.
Time Frame: in 12 weeks of the treatment
Population: Intention-to-treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 528 | 508
Participants | 0 | 0
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p > 0.999, Fisher Exact

5. Secondary Outcome: Presence and Type of Adverse Events (AE).
Description: Based on medical records. Presence and type of adverse events, their severity, relation to investigational drug, outcomes.
Time Frame: in 12 weeks of the treatment
Population: Intention-to-treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Anaferon for Children | Placebo
Number analyzed (Participants) | 528 | 508
Participants
  Mild severity | 65 | 54
  Moderate severity | 4 | 4
Statistical Analysis 1: Comparison: Anaferon for Children vs Placebo; Test type: Superiority; p > 0.999, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse/Serious adverse events were registered during 12 weeks therapy.
Description: Safety evaluation was based on the data from all randomized subjects receiving at least one dose of the study drug (n=1036; Safety population).
Arm/Group | Anaferon for Children | Placebo
All-Cause Mortality (participants affected / at risk) | 0/528 | 0/508
Serious Adverse Events (participants affected / at risk) | 1/528 | 0/508
Other Adverse Events (participants affected / at risk) | 49/528 | 44/508
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anaferon for Children (N=528) | Placebo (N=508)
Partial cramps (Nervous system disorders) | 1 (1) | 0 (0) — Partial epilepsy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anaferon for Children (N=528) | Placebo (N=508)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) — Aphthous stomatitis
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Loose stool
Intestinal dysfunction (Gastrointestinal disorders) | 1 (1) | 0 (0) — Intestinal dysfunction
Teething (Gastrointestinal disorders) | 3 (3) | 1 (1) — Teething
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Vomiting
Functional dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) — Functional dyspepsia
Functional gastrointestinal pathology (Gastrointestinal disorders) | 3 (3) | 1 (1) — Functional gastrointestinal pathology
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Enteritis
Chicken pox (Infections and infestations) | 4 (4) | 8 (8) — Chicken pox
Respiratory viral infection (Infections and infestations) | 3 (3) | 4 (5) — ARVI, rhinopharyngitis
Gastroenteritis caused by norovirus (Infections and infestations) | 0 (0) | 1 (1) — Gastroenteritis caused by norovirus
Herpes on the lips (Infections and infestations) | 0 (0) | 1 (1) — Herpes on the lips
Purulent conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) — Purulent conjunctivitis
Purulent rhinitis (Infections and infestations) | 1 (1) | 1 (1) — Purulent rhinitis
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) — Urinary tract infection
Non-purulent otitis media (Infections and infestations) | 1 (1) | 0 (0) — Non-purulent otitis media
Obstructive bronchitis (Infections and infestations) | 1 (2) | 1 (1) — Obstructive bronchitis
Acute respiratory tract infection (Infections and infestations) | 4 (5) | 4 (4) — Acute respiratory tract infection
Acute nasopharyngitis (Infections and infestations) | 6 (8) | 3 (4) — Acute nasopharyngitis
Acute rhinitis (Infections and infestations) | 0 (0) | 1 (1) — Acute rhinitis
Acute tracheitis (Infections and infestations) | 1 (1) | 2 (2) — Acute tracheitis
Acute pharyngitis (Infections and infestations) | 1 (1) | 1 (1) — Acute pharyngitis
Otitis (Infections and infestations) | 0 (0) | 1 (1) — Otitis
Felon (Infections and infestations) | 0 (0) | 1 (1) — Panaritium
Rhinitis (Infections and infestations) | 2 (2) | 1 (1) — Rhinitis
Rhinosinusitis (Infections and infestations) | 1 (1) | 0 (0) — Rhinosinusitis
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (4) — Rhinopharyngitis
Rotavirus infection (Infections and infestations) | 1 (1) | 1 (1) — Rotavirus infection
Viral otitis media (Infections and infestations) | 0 (0) | 1 (1) — Viral otitis media
Acute otitis media (Infections and infestations) | 1 (1) | 1 (1) — Acute otitis media
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) — Pharyngotonsillitis
Pharyngotracheitis (Infections and infestations) | 1 (1) | 0 (0) — Pharyngotracheitis
Throat hyperemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Throat hyperemia
Runny nose (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) — Runny nose
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Nasal bleeding
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) — Productive cough
Dry cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Dry cough
Allergic rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) — Allergic rash
Allergic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Allergic dermatitis
Skin itch (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Skin itch
Acute allergic urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Acute allergic urticaria
Facial rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash on the skin of the face
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Headache
Partial epilepsy (Nervous system disorders) | 1 (1) | 0 (0) — Partial epilepsy
Fever (General disorders) | 7 (7) | 0 (0) — Fervescence
Stuttering (Psychiatric disorders) | 1 (1) | 0 (0) — Stammering
Foreign body aspiration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Aspiration of a foreign matter

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT03301155/Prot_SAP_000.pdf